CLINICAL TRIAL: NCT01171261
Title: Health Games Research: Advancing Effectiveness of Interactive Games for Health
Brief Title: Testing Health Games for Adolescent Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Greg J. Norman, PhD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RWJ 64439
Record Dates: First submitted 2010-07-23; First posted 2010-07-28 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Sedentary Lifestyle
Keywords: Physical Activity; Sedentary Behavior; Video Games; Exergames
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Jackie Chan Studio Fitness (Experimental): The Jackie Chan Studio Fitness (J-MAT) cartridge includes four types of activities that use a four panel floor mat made of flexible material that functions as the wireless interface game controller. The celebrity actor and choreographer Jackie Chan is the avatar character in the game that demonstrates and guides users in four types of aerobic and anaerobic game modes.
  Interventions: Behavioral: Health Games Field Trial
- XaviX Tennis (Experimental): XaviX Tennis simulates tennis using a tennis racket controller and an infrared sensor to detect speed and timing of the player's swing of the racquet. The Tennis cartridge includes three playing modes. In Tournament Tour players select from eight different characters with different skills and play opponents in a bracketed tournament. In Exhibition mode players choose a computer opponent or play a tennis match with a friend. The Training Games mode includes a) Serving, b) Target Challenge, c) Serve & Finish, and d) Rally Time.
  Interventions: Behavioral: Health Games Field Trial
- XaviX Bowling (Experimental): XaviX Bowling uses a wireless bowling ball game controller to simulate bowling. The cartridge includes three modes. In Regular Game up to four people can select from 8 preset bowlers with different characteristics. In Tournament Mode up to eight people can play. Challenge Games consists of three games called Against the Clock, Moving Pins, and Panel Crusher.
  Interventions: Behavioral: Health Games Field Trial
- XaviX Boxing (Experimental): XaviX Boxing uses boxing gloves as the game controller and allows players to box against five different computer opponents in Championship and Exhibition modes and to practice boxing skills in Exercise mode. Exercise mode includes Punch Fast, Panel Toucher, Punch the Red Ball, and Combination Training.
  Interventions: Behavioral: Health Games Field Trial

INTERVENTIONS:
Behavioral: Health Games Field Trial — There were 4 arms to the intervention in the field trial of this study. Participants were randomized to one of 4 arms or exergame that were manufactured by SSD/Xavix (Shiseido Co. of Japan). Each exergame consisted of a game cartridge, the XavixPort, and game controllers (e.g., tennis racquets, boxing gloves, bowling ball, or floor mat). The XavixPort interfaces the exergame with the participant's television and contains the infrared sensors that track the movement of the game controllers. Each exergame cartridge includes multiple game modes. The four arms/exergames were: XaviX Tennis, The Jackie Chan Studio Fitness (J-MAT), XaviX Bowling, and XaviX Boxing.
  Other Names: Health Games; Exergames

SUMMARY:
This is a RWJF funded study that will apply behavioral choice theory and learning theory principles to 'map' exergames to determine how behavior change principles influence sustained use of health games by adolescents.

DETAILED DESCRIPTION:
This research will assess and map four different exergame sports (bowling, boxing, tennis, and a mat/aerobics) games developed by Xavix for behavioral principles and evaluate how those behavior change principles impact game play sustainability. In the first phase of the study, we mapped and coded video games based on behavior contingencies of antecedents to the behavior, the behavior, and consequences to the behavior. Each of the games and subgames will be categorized as hi fidelity and lo fidelity.

Field Trial A home visit was scheduled for eligible and interested participants and an accelerometer was send to the participant's home to wear for one week prior to the home visit. Participants were randomized to one of four XaviX sports games: tennis, bowling, boxing, or J-mat. Two research assistants visited the participant's home to complete assent and consent forms, install the game on a television in the home, and give an overview on how to play the game. Participants were given a paper game log and instructed to record time spent playing the XaviX games. Participants were asked to play the exergame for as much or as little as they like for the next 4 weeks. The participant and parent completed a baseline survey during the visit. Participants continued to wear the accelerometer during the first week of exergame play and then returned the accelerometer by mail.

During the four weeks of exergame play, participants were contacted by telephone by study staff three times, approximately once a week, to complete short surveys about their game play and attitudes about the exergame, and to address any questions from participants. At week four, participants were mailed an accelerometer and instructed to wear it for seven days. After week four, a second home visit was conducted to collect the game cartridge and system, administer final surveys to the participant and a parent, and distribute the incentive. Participants received $50 for completing all study measurements.

Lab Trial In the lab phase, participants that completed the field trial and were randomized to the bowling, boxing, or J-Mat exergames were eligible to participate in the lab trial. During the lab trial, participants will play two subgames (a hi fidelity and a lo fidelity game) from the game that they were randomized to. Participants also completed a relative reinforcing value (RRV) task to assess reinforcing value of Xavix subgames ranked on theoretical fidelity and exertion. The RRV task is a method to measure the responsiveness of individuals to two or more choices. In the context of competing choice options, the RRV task assesses how much work an individual would be willing to do given increasing response effort to gain access to each option.

ELIGIBILITY:
Inclusion Criteria:

* Are 11 - 15 years
* Provide assent and have a legal guardian that will participate and provide parental permission/consent
* Have a functioning telephone and at least one functioning television

Exclusion Criteria:

* Own another exergame in their home (such as a Wii or Dance Dance Revolution game)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Exergame Sustainability as a Measure of Game Play Over a 4-week Period | 4 weeks
  The amount of game play over a 4-week period was assessed by a self-report paper game play log on which to record the date, start and end time of game play. Participants also indicated the game mode (e.g. challenge games, tournament) and who, if anyone, they played the game with.

SECONDARY OUTCOMES:
Moderate and Vigorous Physical Activity | 4 weeks
  Physical activity was measured by accelerometer before the participant received the XaviX game, during the first week of having the XaviX game in the home, and during the final week that the XaviX game was in the home.
Self-Report of Sedentary Behavior on non-school days | 4 weeks
  Self-reported sedentary time on a typical non-school day was assessed with a previously developed measure survey adapted from Robinson (1999). Participants were asked how much time they spent doing the following sedentary behaviors: (a) watching TV (including videos on VCR/DVD); (b) playing computer or video games (like Nintendo or Sega); (c) using the internet, emailing or other electronic media for leisure; (d) doing homework; (e) reading a book or magazine (not for school); (f) riding in a car, bus, etc.
Attitudes about Exergames | 4 weeks
  Self-report of attitudes about exergames and the XaviX system were assessed through a 12-item scale on feelings about exergames, a price point question for the XaviX system and XaviX game cartridges, a survey on participants' experience with the XaviX system and game and why they would play XaviX in the future.
Motivation to Play Exergames | 4 weeks
  A Motivation for Exergame Play Inventory was developed to assess motivation for exergame play.

CONTACTS AND LOCATIONS:
Overall Officials: Greg J Norman, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD, Atkinson Hall, 3rd Floor, La Jolla, California, United States